CLINICAL TRIAL: NCT05653037
Title: A Randomized, Single-blind, Placebo-Controlled Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses of Subcutaneously Administered RBD4059 in Healthy Subjects
Brief Title: A Single Ascending Doses Phase I Study to Evaluate the Safety and Pharmacokinetics of RBD4059 in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Ribo Life Science Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: RBFI1101
Record Dates: First submitted 2022-11-21; First posted 2022-12-16 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RBD4059 SAD experimental group (Experimental): Subjects in SAD experimental groups will receive a single subcutaneous injection of RBD4059 on Day 1.
  Interventions: Drug: RBD4059
- Placebo SAD group (Placebo Comparator): Subjects in SAD placebo groups will receive a single subcutaneous injection of placebo on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RBD4059 — Subcutaneously Administered RBD4059 in Healthy Subjects.
  Arms: RBD4059 SAD experimental group
Drug: Placebo — Subcutaneously Administered Placebo in Healthys Subject.
  Arms: Placebo SAD group

SUMMARY:
This is a Randomized, Single-blind, Placebo-Controlled Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses of Subcutaneously Administered RBD4059 in Healthy Subjects. The study will be performed in single ascending dose (SAD) phase in healthy subjects. The decision to escalate to subsequent dose levels will be made by the SRC based on the review of all available safety information and PK/PD data in each cohort.

RBD4059, a GalNAc conjugated siRNA, is an FXI-targeted new molecular entity independently developed by Ribo using its proprietary siRNA delivery system - RIBO-GalSTARTM.

DETAILED DESCRIPTION:
RBD4059, a GalNAc conjugated siRNA, is an FXI-targeted new molecular entity independently developed by Ribo using its proprietary siRNA delivery system - RIBO-GalSTARTM. As a GalNAc-based liver targeting delivery system, RIBO-GalSTARTM incorporates a unique technology for the delivery of oligonucleotide therapeutics for various targets and indications associated with the liver, thus enabling highly specific and highly durable enrichment of the siRNA in hepatocytes, the primary source of FXI. RBD4059 is, therefore, proposed to be a novel effective and durable antithrombotic treatment, with low bleeding risk via inhibition of FXI activity and prolongation of APTT.

ELIGIBILITY:
Inclusion Criteria:

* Male and female (non-childbearing potential only), aged 18 to 65 years, inclusive.
* Body mass index (BMI) between 18 and 32 kg/m2, inclusive.
* APTT, Prothrombin time(PT), INR, thrombin time (TT)，FXI activity must be within the normal reference range (as per the local laboratory reference range) at screening .
* Adequate complete blood counts (CBCs) and platelet are within the normal reference range (If CBCs are outside the reference range, unless not clinically significant determined by the Investigator ).
* Healthy as determined by pre-study medical history, vital signs, physical examination, clinical laboratory assessments, and 12-lead electrocardiogram (ECG).
* Subjects who are willing to cooperate with the study staff, comply with the study requirements, complete the study according to the relevant procedures specified in the protocol, and correctly understand and sign the informed consent form in writing.

Exclusion Criteria:

* Any uncontrolled or serious disease that may interfere with participation in the clinical study and/or put the subject at significant risk (according to Investigator's judgment) if he/she participates in the clinical study.
* History or presence of cardiovascular disease (including peripheral artery and cerebrovascular disease).
* Systolic blood pressure (SBP) is less than 90 or greater than 140 mmHg and/or diastolic blood pressure (DBP) is less than 40 or greater than 90 mmHg after 10 minutes of supine rest, unless determined by the Investigator to be not clinically significant.
* Diagnosis of diabetes mellitus, history of gestational diabetes that is fully resolved is not permitted.
* Any conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study.

Note: additional inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Related Adverse Events as Assessed by CTCAE v5.0 | SAD: Up to Day 169 ;

SECONDARY OUTCOMES:
To characterize the pharmacokinetics (PK) of RBD4059 in healthy subjects:Cmax | Up to 48 hours post-dose
To characterize the pharmacokinetics (PK) of RBD4059 in healthy subjects:Tmax | Up to 48 hours post-dose
To characterize the pharmacokinetics (PK) of RBD4059 in healthy subjects:AUC0-t | Up to 48 hours post-dose
To characterize the pharmacokinetics (PK) of RBD4059 in healthy subjects:AUC0-inf | Up to 48 hours post-dose
To characterize the pharmacokinetics (PK) of RBD4059 in healthy subjects:t1/2 | Up to 48 hours post-dose
To characterize the pharmacokinetics (PK) of RBD4059 in healthy subjects:MRT | Up to 48 hours post-dose
To characterize the pharmacokinetics (PK) of RBD4059 in healthy subjects:λz | Up to 48 hours post-dose
To characterize the pharmacokinetics (PK) of RBD4059 in healthy subjects:CL/F | Up to 48 hours post-dose
To characterize the pharmacokinetics (PK) of RBD4059 in healthy subjects:Vz | Up to 48 hours post-dose
To evaluate the pharmacodynamics (PD) effect of RBD4059 on levels of Coagulation factor XI (FXI) antigen in healthy subjects. | SAD: Up to Day 169 ;
To evaluate the pharmacodynamics (PD) effect of RBD4059 on levels of FXI activity in healthy subjects. | SAD: Up to Day 169 ;
To evaluate the pharmacodynamics (PD) effect of RBD4059 on levels of Activated partial thromboplastin time (APTT) in healthy subjects. | SAD: Up to Day 169 ;

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Pharm Pty Limited, Brisbane, Australia